CLINICAL TRIAL: NCT04577898
Title: A Randomized, Blinded Evaluator, No-treatment Control, Multicenter, Prospective Clinical Study of RHA® Redensity Eye for the Treatment of Moderate to Severe Tissue Volume Deficiencies in the Infraorbital Regions
Brief Title: RHA® Redensity Eye Versus No-treatment for the Infra-Orbital Hollows
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teoxane SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TEO-RHA-1902
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Infra-orbital Hollows; Tear-trough Deformity; Wrinkle
Keywords: Dermal Filler; Hyaluronic acid; Infra-orbital Hollows; Tear-trough deformity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- RHA® Redensity Eye Group (Experimental): RHA® Redensity Eye is injected from the sub-dermis to the periosteum in the infraorbital hollow.
  Up to 1.0 mL per eye at each treatment (max: 2.0 mL per treatment). No touch-up treatment provided.
  Interventions: Device: RHA® Redensity Eye
- No-Treatment Control First, Then RHA Redensity Eye Treatment Group (No Intervention): During Phase 1a, participants from No-treatment control group do not receive treatment. Primary endpoint assessments are done at Week 12. Once all evaluations applicable for Primary Endpoint at Week 12 are completed, subjects proceed directly to Phase 1b (on the same day).
  Phase 1b is only applicable to subjects initially randomly assigned to the No-treatment control group.
  Phase 1b: Subjects receive their initial treatment with RHA® Redensity Eye at Visit 1b.
  Subjects follow the same schedule as those initially randomly assigned to the RHA® Redensity Eye group: RHA® Redensity Eye is administered on the same day (Visit 1b). Subjects come to the site 12 weeks after their initial treatment.
  RHA® Redensity Eye is injected from the sub-dermis to the periosteum in the infraorbital hollow.
  Up to 1.0 mL per eye at each treatment (max: 2.0 mL per treatment). No touch-up treatment provided.

INTERVENTIONS:
Device: RHA® Redensity Eye — A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of streptococcus zooepidemicus, formulated to a concentration of 15 mg/g and 0.3% w/w lidocaine in a physiologic buffer.
  Arms: RHA® Redensity Eye Group

SUMMARY:
This is a multicenter, blinded evaluator, randomized, prospective, no treatment control clinical study to identify whether RHA® Redensity Eye (*) is superior to no treatment for the correction of moderate to severe tissue volume deficiencies in the infraorbital regions.

The study will include at least 20% of subjects with Fitzpatrick skin types IV-VI.

The Treating Investigator (TI) and the Blinded Live Evaluator (BLE) will evaluate the subject's infraorbital hollows independently of each other using the Teoxane Infraorbital Hollows Scale (TIOHS) at Screening (Visit 1) for eligibility.

If the subject is eligible, the BLE's assessment will be used for the Baseline of the primary endpoint.

Enrolled subjects will be randomly assigned in a ratio of 3:1 at Screening (Visit 1) to receive RHA® Redensity Eye or to receive no treatment (No-treatment control group).

Subjects receiving RHA® Redensity Eye will be further divided by the method of administration (i.e. injection with a 30G ½" needle or 25G 1 ½" cannula), which will be defined for each site at the beginning of the study. Site selection will aim to achieve approximately 1:1 distribution between the administration method subgroups. The BLE will be blinded to the study groups (RHA® Redensity Eye group or No treatment control group).

For subjects randomly assigned to RHA® Redensity Eye group, the study will be conducted in 2 Phases - Phase 1a and Phase 2.

For subjects randomly assigned to No-treatment control group, the study will be conducted in 3 Phases - Phase 1a, Phase 1b and Phase 2.

The Phase 1b is not applicable for the subject assigned to the RHA® Redensity Eye group.

(*): TEO-RHA-1902 was conducted with RHA® Redensity Eye Lido, that contains Lidocaine.

DETAILED DESCRIPTION:
Phase 1a:

Subjects who will be randomly assigned to the RHA® Redensity Eye group at Screening will receive their injection at Visit 1. Subjects will come to the site 12 weeks (primary endpoint) after the initial treatment. Afterwards, subjects will proceed directly to Phase 2.

Subjects randomly assigned to the No-treatment control group at Screening will receive no treatment in Phase 1a of the study. They will come to the site 12 weeks (primary endpoint) after randomization. After completing all assessments, subjects will immediately begin Phase 1b (Visit 1b is on the same day as Visit at Week 12) and will receive their initial treatment with RHA® Redensity Eye.

Phase 1b:

Phase 1b is only applicable to subjects initially randomly assigned to the No-treatment control group. Once all evaluations applicable for Visit at Week 12 are completed, subjects will proceed directly to Visit 1b (on the same day). Evaluations completed at Week 12 will be used for Visit 1b and will become the new Baseline for Phase 1b.

Subjects will receive their initial treatment with RHA® Redensity Eye at Visit 1b.

Subjects will follow the same schedule as those initially randomly assigned to the RHA® Redensity Eye group: RHA® Redensity Eye will be administered on the same day (Visit 1b). Subjects will come to the site 12 weeks after their initial treatment. Afterwards, subjects will proceed to Phase 2.

Phase 2 and Exit visit:

Phase 2 will occur 12 weeks after receiving initial treatment with RHA® Redensity Eye for subjects in the RHA® Redensity Eye group and the No-treatment control group (after Phase 1b).

All these subjects will come to the site 24 weeks, and 52 weeks after their initial treatment. All subjects will be followed for 52 weeks after their initial treatment with RHA® Redensity Eye.

Subjects will be offered retreatment (52 weeks after their initial treatment). Retreatment will be administered if the TI deems it to be appropriate and the subject agrees. If the subject does not receive retreatment, Visit at 52 weeks after initial treatment will become the Exit visit.

If the subject receives retreatment, the subjects will come to the site 12 weeks after retreatment for follow-up and safety assessments. This will be the Exit visit.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female of any race, 22 years of age or older
* Infra-orbital Hollows of grade 2 to 3 on the TIOHS (ranging from 0 to 4) who is seeking treatment of moderate to severe tissue volume deficiencies in the infra-orbital region (realistic and achievable as per TI opinion). Bilateral symmetry is not required. If the assessments of the TI and the BLE are the same or differ by exactly 1 point on the scale, this difference is considered acceptable. If the subject is eligible, the BLE's assessment will be used for the Baseline for the primary endpoint. If the TI and the BLE do not agree on eligibility, or if their assessments differ by 2 points or more on the scale, the subject will not be eligible.
* Willing to abstain from facial aesthetic procedures/therapies that could interfere with study evaluations
* Able to follow study instructions and complete all required visits.
* Sign the IRB-approved ICF, Photographic Release Form and the Authorization for Use and release of Health and Research Study Information (HIPAA) form prior to any study- related procedures being performed.

Exclusion Criteria:

* Female subjects that are pregnant, breast-feeding or of childbearing potential and not practicing reliable birth control
* Known hypersensitivity/allergy to any component of the study devices
* Clinically significant active skin disease within 6 months
* Has a history of or currently has an auto-immune disease.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2025-02-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - United States, California, Encino, California
  - United States, Santa Monica, Santa Monica, California
  - United States, Florida, Coral Gables, Florida
  - United States, Illinois, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Groups:
- RHA Redensity Eye Group: Phase 1a RHA® Redensity Eye is injected from the sub-dermis to the periosteum in the infraorbital hollow.
  Up to 1.0 mL per eye at each treatment (max: 2.0 mL per treatment). No touch-up treatment provided.
  RHA® Redensity Eye: A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of streptococcus zooepidemicus, formulated to a concentration of 15 mg/g and 0.3% w/w lidocaine in a physiologic buffer.
- No-Treatment Control First, Then RHA Redensity Eye Treatment Group: During Phase 1a, participants from No-treatment control group do not receive treatment. Primary endpoint assessments are done at Week 12. Once all evaluations applicable for Primary Endpoint at Week 12 are completed, subjects proceed directly to Phase 1b (on the same day).
  Phase 1b is only applicable to subjects initially randomly assigned to the No-treatment control group.
  Phase 1b: Subjects receive their initial treatment with RHA® Redensity Eye at Visit 1b.
  Subjects follow the same schedule as those initially randomly assigned to the RHA® Redensity Eye group: RHA® Redensity Eye is administered on the same day (Visit 1b). Subjects come to the site 12 weeks after their initial treatment.
  RHA® Redensity Eye is injected from the sub-dermis to the periosteum in the infraorbital hollow.
  Up to 1.0 mL per eye at each treatment (max: 2.0 mL per treatment). No touch-up treatment provided.
  RHA® Redensity Eye: A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of streptococcus zooepidemicus, formulated to a concentration of 15 mg/g and 0.3% w/w lidocaine in a physiologic buffer.
- Pooled Safety Assessment: All Participants: Phases 1a, 1b and 2 Pooled data (i.e., after the No-Treatment group received RHA® Redensity Eye after primary endpoint at Week 12, data from both treatment groups were pooled) were used to assess the overall safety of RHA® Redensity Eye as well as effectiveness of RHA® Redensity Eye over time up to 52 weeks after treatment and 12 weeks following retreatment.
  RHA® Redensity Eye is injected from the sub-dermis to the periosteum in the infraorbital hollow.
  Up to 1.0 mL per eye at each treatment (max: 2.0 mL per treatment). No touch-up treatment provided.
  RHA® Redensity Eye: A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of streptococcus zooepidemicus, formulated to a concentration of 15 mg/g and 0.3% w/w lidocaine in a physiologic buffer.
Period: Period 1: Phase 1a
Arm/Group | RHA Redensity Eye Group | No-Treatment Control First, Then RHA Redensity Eye Treatment Group | Pooled Safety Assessment: All Participants
Started (ITT Population) | 183 | 65 | 0
ITT Population | 183 | 65 | 0
PP Population | 167 | 51 | 0
Completed | 173 | 52 | 0
Not Completed | 10 | 13 | 0
Period: Period 2: Phase 1b
Arm/Group | RHA Redensity Eye Group | No-Treatment Control First, Then RHA Redensity Eye Treatment Group | Pooled Safety Assessment: All Participants
Started (SAFT - ITT Population) | 0 | 50 | 0
SAFT - ITT Population | 0 | 50 | 0
PP Population | 0 | 50 | 0
Completed | 0 | 48 | 0
Not Completed | 0 | 2 | 0
Period: Period 3: Phase 2
Arm/Group | RHA Redensity Eye Group | No-Treatment Control First, Then RHA Redensity Eye Treatment Group | Pooled Safety Assessment: All Participants
Started | 0 | 0 | 233
SAFT - ITT Population | 0 | 0 | 233
PP Population | 0 | 0 | 217
Completed | 0 | 0 | 203
Not Completed | 0 | 0 | 30

BASELINE CHARACTERISTICS:
Groups:
- RHA Redensity Eye Group: Phase 1a RHA® Redensity Eye is injected from the sub-dermis to the periosteum in the infraorbital hollow.
  RHA® Redensity Eye is injected from the sub-dermis to the periosteum in the infraorbital hollow.
  Up to 1.0 mL per eye at each treatment (max: 2.0 mL per treatment). No touch-up treatment provided.
  RHA® Redensity Eye: A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of streptococcus zooepidemicus, formulated to a concentration of 15 mg/g and 0.3% w/w lidocaine in a physiologic buffer.
- Total: Total of all reporting groups
Arm/Group | RHA Redensity Eye Group | No-Treatment Control First, Then RHA Redensity Eye Treatment Group | Total
Number analyzed (Participants) | 183 | 65 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (10.65) | 48.2 (11.11) | 49.5 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 60 | 220
  Male | 23 | 5 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 6 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 16 | 5 | 21
  White | 151 | 58 | 209
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 183 | 65 | 248
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick skin type as determined by the Treating Investigator on the skin tone scale developed to classify skin coloring and response to ultraviolet (UV) radiation. The scale contains 6 grades:
  I: Pale white skin; Always burns, does not tan. II: Fair skin; Burns easily, tans poorly. III: Darker white skin; Tans after initial burn. IV: Light brown skin; Burns minimally, tans easily. V: Brown skin; Rarely burns, tans darkly easily. VI: Dark brown or black skin; Never burns, always tans darkly.
  Participants
    Type I-III | 119 | 42 | 161
    Type IV-VI | 64 | 23 | 87

OUTCOME MEASURES:

1. Primary Outcome: Change of 1 Point From Baseline in Infra-Orbital Hollows Severity Rated by the Blinded Live Evaluator (BLE) at Week 12 After Last Treatment, Using the TIOHS - Phase 1a
Description: The TIOHS is a validated 5-point scale for assessing Infra-orbital hollows severity. Possible scores range from 0 (Absent) to 4 (Very Severe).
  Change = (Week 12 - Baseline score). A TIOHS change of 1-grade will be considered clinically significant. Phase 1a: Subjects are randomly assigned to the RHA® Redensity Eye group or to the to the No-treatment control group, and come to the site 12 weeks (primary endpoint) after randomization.
Time Frame: Period 1 - Phase 1a: Week 12 after last treatment
Population: Period 1: Phase 1a - Primary endpoint on the ITT population
Measure: Number; unit: percentage of responders
Arm/Group | RHA Redensity Eye Group | No-Treatment Control First, Then RHA Redensity Eye Treatment Group
Number analyzed (Participants) | 183 | 65
percentage of responders | 79 | 9

2. Primary Outcome: The Modified FACE-Q "Appearance of Lower Eyelids" Change From Baseline Score for Subjects Treated With RHA® Redensity at Week 12 After Last Treatment - Phase 1a
Description: The FACE-Q measures the experience and outcomes of aesthetic facial procedures from the patient's perspective.
  The modified FACE-Q questionnaire is composed of 4 questions with a score linked to answers (1 being "Not at all" and 4 being "Extremely").
  To calculate the FACE-Q score, outcomes from all 4 questions were pooled, data were transformed so that higher scores reflected a superior (positive) outcome, and adapted to a scale of 100 units (i.e. worst/lowest score = 0, best/highest score = 100).
  Phase 1a: Subjects are randomly assigned to the RHA® Redensity Eye group or to the to the No-treatment control group, and come to the site 12 weeks (primary endpoint) after randomization.
Time Frame: Period 1 - Phase 1a: Change from Baseline at Week 12 after last treatment
Population: Period 1 -ITT Population
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- RHA® Redensity Eye Group: Phase 1a RHA® Redensity Eye is injected from the sub-dermis to the periosteum in the infraorbital hollow.
  Up to 1.0 mL per eye at each treatment (max: 2.0 mL per treatment). No touch-up treatment provided.
  RHA® Redensity Eye: A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of streptococcus zooepidemicus, formulated to a concentration of 15 mg/g and 0.3% w/w lidocaine in a physiologic buffer.
Arm/Group | RHA® Redensity Eye Group | No-Treatment Control First, Then RHA Redensity Eye Treatment Group
Number analyzed (Participants) | 183 | 65
score on a scale | 37.5 (27.04) | -4.1 (17.48)

3. Secondary Outcome: Number of Subjects Who Scored Themselves Either "Much Improved" or "Improved" on Global Aesthetic Improvement (GAI) Scale by the Subject at Weeks 12, 24, 52 After Last Treatment and at Week 12 After Retreatment - Phase 2
Description: The Global Aesthetic Improvement (GAI) is a subjective, balanced, 5-point dynamic scale assessing cosmetic improvement.
  Possible scores range from "much improved", "improved", "no change", "worse", to "much worse".
  The GAI will be assessed using the pre-injection baseline photograph. Phase 3 - Phase 2: Subjects from No-Treatment group receive their treatment with RHA® Redensity Eye following primary endpoint assessment, and enter into Phase 2. Phase 2 occur 12 weeks after receiving initial treatment with RHA® Redensity Eye for subjects in the RHA® Redensity Eye group and the No-treatment control group, data are pooled for analysis.
Time Frame: Period 3: Phase 2 - ITT population - Weeks 12, 24, 52 after last treatment and at Week 12 after retreatment.
Population: Phase 2 - ITT population - Weeks 12, 24, 52 after last treatment and at Week 12 after retreatment.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Population: All Participants: Phase 2 Pooled data (i.e., after the No-Treatment group received RHA® Redensity Eye after primary endpoint at Week 12, data from both treatment groups were pooled) were used to assess the overall safety of RHA® Redensity Eye as well as effectiveness of RHA® Redensity Eye over time up to 52 weeks after treatment and 12 weeks following retreatment.
Arm/Group | Pooled Population: All Participants
Number analyzed (Participants) | 233
Participants
  Week 12 after last treatment: number analyzed (Participants) | 221
  Week 12 after last treatment | 197
  Week 24 after last treatment: number analyzed (Participants) | 213
  Week 24 after last treatment | 176
  Week 52 after last treatment: number analyzed (Participants) | 205
  Week 52 after last treatment | 135
  Week 12 after retreatment: number analyzed (Participants) | 99
  Week 12 after retreatment | 89

4. Secondary Outcome: Number of Subjects Scored Themselves Either "Much Improved" or "Improved" on Global Aesthetic Improvement (GAI) Scale by the Blinded Live Evaluator (BLE) at Weeks 12, 24, 52 After Last Treatment and at Week 12 After Retreatment - Phase 2
Description: The Global Aesthetic Improvement (GAI) is a subjective, balanced, 5-point dynamic scale assessing cosmetic improvement.
  Possible scores range from "much improved", "improved", "no change", "worse", to "much worse".
  The GAI will be assessed using the pre-injection baseline photograph. Phase 2: Subjects from No-Treatment group receive their teatment with RHA® Redensity Eye following primary endpoint assessment, and enter into Phase 2. Phase 2 occur 12 weeks after receiving initial treatment with RHA® Redensity Eye for subjects in the RHA® Redensity Eye group and the No-treatment control group, data are pooled for analysis.
Time Frame: Period 3 - Phase 2 - ITT population - Weeks 12, 24, 52 after last treatment and at Week 12 after retreatment.
Population: Period 3 -Phase 2 - ITT population - Weeks 12, 24, 52 after last treatment and at Week 12 after retreatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Population: All Participants
Number analyzed (Participants) | 233
Participants
  Week 12 after last treatment: number analyzed (Participants) | 221
  Week 12 after last treatment | 205
  Week 24 after last treatment: number analyzed (Participants) | 213
  Week 24 after last treatment | 187
  Week 52 after last treatment: number analyzed (Participants) | 205
  Week 52 after last treatment | 152
  Week 12 after retreatment: number analyzed (Participants) | 99
  Week 12 after retreatment | 90

5. Secondary Outcome: Number of Subjects "Satisfied" or "Very Satisfied" With Study Treatment Using the Subject Satisfaction Scale at Weeks 12, 24, 52 After Initial Treatment and at Week 12 After Retreatment - Phase 2
Description: The Subject Satisfaction Scale is a subjective, balanced, 5-point scale assessing subject satisfaction with study treatment. Possible scores range from with 1 (very satisfied) to 5 (very dissatisfied).
  Period 3 - Phase 2: Subjects from No-Treatment group receive their teatment with RHA® Redensity Eye following primary endpoint assessment, and enter into Phase 2. Phase 2 occur 12 weeks after receiving initial treatment with RHA® Redensity Eye for subjects in the RHA® Redensity Eye group and the No-treatment control group, data are pooled for analysis.
Time Frame: Period 3: Phase 2 - ITT population - Weeks 12, 24, 52 after initial treatment and at Week 12 after retreatment.
Population: Period 3 - Phase 2 - ITT population - Weeks 12, 24, 52 after last treatment and at Week 12 after retreatment.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Population : All Participants: Phase 2 Pooled data (i.e., after the No-Treatment group received RHA® Redensity Eye after primary endpoint at Week 12, data from both treatment groups were pooled) were used to assess the overall safety of RHA® Redensity Eye as well as effectiveness of RHA® Redensity Eye over time up to 52 weeks after treatment and 12 weeks following retreatment.
Arm/Group | Pooled Population : All Participants
Number analyzed (Participants) | 233
Participants
  Week 12 after last treatment: number analyzed (Participants) | 220
  Week 12 after last treatment | 174
  Week 24 after last treatment: number analyzed (Participants) | 213
  Week 24 after last treatment | 154
  Week 52 after last treatment: number analyzed (Participants) | 205
  Week 52 after last treatment | 133
  Week 12 after retreatment: number analyzed (Participants) | 99
  Week 12 after retreatment | 83

6. Secondary Outcome: Change of 1 Point From Baseline in Infra-Orbital Hollows Severity Rated by the Blinded Live Evaluator (BLE) at Weeks 12, 24, 52 After Initial Treatment and at Week 12 After Retreatment Using the TIOHS - Phase 2
Description: The TIOHS is a validated 5-point scale for assessing Infra-orbital hollows severity. Possible scores range from 0 (Absent) to 4 (Very Severe).
  Period 3 - Phase 2: Subjects from No-Treatment group receive their teatment with RHA® Redensity Eye following primary endpoint assessment, and enter into Phase 2. Phase 2 occur 12 weeks after receiving initial treatment with RHA® Redensity Eye for subjects in the RHA® Redensity Eye group and the No-treatment control group, data are pooled for analysis.
Time Frame: Period 3: Phase 2 - ITT population - Weeks 12, 24, 52 after initial treatment and at Week 12 after retreatment.
Population: Period 3: Phase 2 - ITT population - Weeks 12, 24, 52 after last treatment and at Week 12 after retreatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Population: All Participants
Number analyzed (Participants) | 233
Participants
  Week 12 after last treatment: number analyzed (Participants) | 221
  Week 12 after last treatment | 173
  Week 24 after last treatment: number analyzed (Participants) | 213
  Week 24 after last treatment | 159
  Week 52 after last treatment: number analyzed (Participants) | 205
  Week 52 after last treatment | 124
  Week 12 after retreatment: number analyzed (Participants) | 99
  Week 12 after retreatment | 79

7. Secondary Outcome: Subject's Perception of Treatment Effectiveness as Per the "Appearance of Lower Eyelids " FACE-Q Scale Questionnaire at Baseline, Weeks 12, 24, 52 After Initial Treatment and at Week 12 After Retreatment - Phase 2
Description: The FACE-Q measures the experience and outcomes of aesthetic facial procedures from the patient's perspective.
  The FACE-Q questionnaire is composed of 7 questions with a score linked to answers (1 being "Not at all" and 4 being "Extremely").
  To calculate the FACE-Q score, outcomes from all 7 questions were pooled, data were transformed so that higher scores reflected a superior (positive) outcome, and adapted to a scale of 100 units (i.e. worst/lowest score = 0, best/highest score = 100).
  Period 3 - Phase 2: Subjects from No-Treatment group receive their teatment with RHA® Redensity Eye following primary endpoint assessment, and enter into Phase 2. Phase 2 occur 12 weeks after receiving initial treatment with RHA® Redensity Eye for subjects in the RHA® Redensity Eye group and the No-treatment control group, data are pooled for analysis.
Time Frame: Period 3: Phase 2 - ITT population - Change from Baseline at Weeks 12, 24, 52 after initial treatment and at Week 12 after retreatment.
Population: Period 3:Phase 2 - ITT population - Weeks 12, 24, 52 after last treatment and at Week 12 after retreatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pooled Population: All Participants
Number analyzed (Participants) | 233
score on a scale
  Week 12 after last treatment: number analyzed (Participants) | 221
  Week 12 after last treatment | 26.6 (24.77)
  Week 24 after last treatment: number analyzed (Participants) | 213
  Week 24 after last treatment | 23.2 (24.09)
  Week 52 after last treatment: number analyzed (Participants) | 205
  Week 52 after last treatment | 15.1 (23.97)
  Week 12 after retreatment: number analyzed (Participants) | 99
  Week 12 after retreatment | 30.7 (25.52)

ADVERSE EVENTS:
Time Frame: 52 to 64 (for patients receiving re-treatment) weeks
Groups:
- Pooled Safety Assessment: Phases 1a, 1b and 2 Pooled data (i.e., after the No-Treatment group received RHA® Redensity Eye after primary endpoint at Week 12, data from both treatment groups were pooled) were used to assess the overall safety of RHA® Redensity Eye as well as effectiveness of RHA® Redensity Eye over time up to 52 weeks after treatment and 12 weeks following retreatment.
  RHA® Redensity Eye is injected from the sub-dermis to the periosteum in the infraorbital hollow.
  Up to 1.0 mL per eye at each treatment (max: 2.0 mL per treatment). No touch-up treatment provided.
  RHA® Redensity Eye: A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of streptococcus zooepidemicus, formulated to a concentration of 15 mg/g and 0.3% w/w lidocaine in a physiologic buffer.
  For the pooled population, of the 65 subjects in the No-Treatment group, 13 did not reach Week 12 to crossover and receive RHA Redensity® Eye Lido treatment and 2 of the 50 who reached Week 12 did not receive treatment at that visit. Therefore, there were 233 subjects as part of SAFT for the pooled data set
Arm/Group | RHA Redensity Eye Group | No-Treatment Control First, Then RHA Redensity Eye Treatment Group | Pooled Safety Assessment
All-Cause Mortality (participants affected / at risk) | 0/183 | 0/65 | 0/233
Serious Adverse Events (participants affected / at risk) | 0/183 | 0/65 | 2/233
Other Adverse Events (participants affected / at risk) | 28/183 | 0/65 | 30/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RHA Redensity Eye Group (N=183) | No-Treatment Control First, Then RHA Redensity Eye Treatment Group (N=65) | Pooled Safety Assessment (N=233)
Cholecystitis Acute (Hepatobiliary disorders) | NA | NA | 1 (1)
Cellulitis (Infections and infestations) | NA | NA | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RHA Redensity Eye Group (N=183) | No-Treatment Control First, Then RHA Redensity Eye Treatment Group (N=65) | Pooled Safety Assessment (N=233)
Injection Site Discolouration (General disorders) | 10 | 0 | 12
Injection Site Mass (General disorders) | 6 | 0 | 9
Injection Site Swelling (General disorders) | 3 | 0 | 9
Headache (Nervous system disorders) | 12 | 0 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-04-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT04577898/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT04577898/SAP_001.pdf